CLINICAL TRIAL: NCT00855439
Title: A Single-center,Proof of Concept,Randomized,Controlled Parallel Group Clinical Trial of the Effects of Exenatide vs. a Long Acting Insulin Analog to Evaluate the Efficacy of Exenatide in Patients With Diabetic Neuropathy and Type 2 Diabetes
Brief Title: Evaluation of Exenatide in Patients With Diabetic Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Amylin Pharmaceuticals, LLC. (Industry); Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Rodica Pop-Busui, Assistant Professor of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H80-US-X012
Record Dates: First submitted 2009-03-03; First posted 2009-03-04 (Estimated); Results first posted 2015-05-12 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-01

CONDITIONS: Type 2 Diabetes Mellitus; Diabetic Peripheral Neuropathy
Keywords: Diabetes; Neuropathy; Glucose; Control; Peripheral; Autonomic
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Exenatide; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exenatide (Experimental): Subjects will take exenatide by subcutaneous injection twice daily for 18 months
  Interventions: Drug: Exenatide
- glargine (Active Comparator): Subjects will take 1 daily injection of insulin glargine for 18 months.
  Interventions: Drug: Glargine

INTERVENTIONS:
Drug: Exenatide — Exenatide is given according to current FDA prescribing guidelines. Exenatide and other diabetes medications will be titrated in order to achieve optimal blood glucose levels
  Other Names: Byetta
  Arms: Exenatide
Drug: Glargine — Subjects will take 1 daily injection of insulin glargine in manner consistent with current prescribing guidelines. Glargine and other diabetes medications will be adjusted to achieve optimal levels of blood sugar control
  Other Names: Lantus
  Arms: glargine

SUMMARY:
This study will look at whether or not the medication exenatide improves signs and symptoms of diabetic peripheral neuropathy in people with type 2 diabetes and mild to moderate diabetic peripheral neuropathy.

DETAILED DESCRIPTION:
This study will look at the effects of the medication exenatide on peripheral neuropathy in people with type 2 diabetes. Exenatide (trade name, BYETTA®) is an injectable medication used by people with type 2 diabetes to control blood sugar. Peripheral neuropathy is a complication of diabetes that can cause symptoms such as numbness, tingling or burning sensations in the feet and hands. Controlling blood sugars levels in type 2 diabetes is thought to prevent, delay or improve the damage to the nerve fibers that causes peripheral neuropathy. There is also some evidence that exenatide may have additional beneficial effects on the peripheral nerves, beyond the benefits of blood sugar control alone. In this study, about half of the participants will take exenatide by injection twice daily and the other half will take insulin glargine (Lantus®) by injection once daily. Both groups are expected to have similar improvement in blood sugar control. This study will show whether exenatide has beneficial effects on neuropathy beyond the benefits of better blood sugar control alone.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes treated with one or more oral agents
* Persistent fasting glucose > 140 mg/dl or HbA1c > 7%
* Stable and maximally effective doses of one or more oral agents for 3 months
* Presence of diabetic peripheral neuropathy
* Age between 18 and 70 years
* No risk factors or other causes of neuropathy
* Willingness and capacity to sign the Institutional Review Board approved consent form and cooperate with the medical procedures for study duration

Exclusion Criteria:

* Nursing mothers or pregnant women
* A history of previous kidney, pancreas or cardiac transplantation
* A past history of neuropathy (independent of diabetes) or with a disease known to be associated with neuropathy (e.g., hepatitis C, end stage renal disease, lupus)
* Amputation of any part of either lower extremity for any reason or traumatic loss of any part of either lower extremity or congenital absence or severe deformity of lower extremity
* HbA1c > 10%
* Participation in an experimental medication trial within 3 months of starting the study.
* Undergoing therapy for malignant disease other than basal- or squamous cell carcinoma
* Requiring long-term glucocorticoid therapy
* Inability or unwillingness to comply with the protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2008-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodica Pop-Busui, MD, PhD, Principal Investigator — University of Michigan
Locations (1):
- The University of Michigan Health System, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jaiswal M, Martin CL, Brown MB, Callaghan B, Albers JW, Feldman EL, Pop-Busui R. Effects of exenatide on measures of diabetic neuropathy in subjects with type 2 diabetes: results from an 18-month proof-of-concept open-label randomized study. J Diabetes Complications. 2015 Nov-Dec;29(8):1287-94. doi: 10.1016/j.jdiacomp.2015.07.013. Epub 2015 Jul 17. PMID 26264399

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Date of first patient randomized to treatment:10/29/2008 Date of last patient randomized to treatment:12/07/2012
Pre-assignment Details: After obtaining written informed consent, participants were asked to provide medical history. A physical examination was performed, with specific focus on signs and symptoms of peripheral neuropathy. Baseline labs were obtained. Eligible subjects were invited for a baseline visit at which detailed neurologic assessment were done.
Period: Overall Study
Arm/Group | Exenatide | Glargine
Started | 22 | 24
Completed | 19 | 24
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Pregnancy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exenatide | Glargine | Total
Number analyzed (Participants) | 22 | 24 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 20 | 36
  >=65 years | 6 | 4 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (13) | 54 (9) | 53 (10)
Gender [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 13 | 13 | 26
Region of Enrollment [Number; unit: participants]
  United States | 22 | 24 | 46

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Clinical Neuropathy (CCN)
Description: CCN was defined by a composite score comprised of at least two positive responses among symptoms, sensory signs, or absent or hypoactive reflexes consistent with a distal symmetrical polyneuropathy (16), and at least one abnormal nerve conduction study result in two anatomically distinct nerves, e.g. the sural sensory and peroneal motor nerves (defined as a amplitude < 5 μV and a conduction velocity < 40 m/sec for the sural nerve and an amplitude < 2.5 μV and a conduction velocity < 40 m/sec for the peroneal nerve).
Time Frame: 18 Months
Measure: Number; unit: participants
Arm/Group | Exenatide | Glargine
Number analyzed (Participants) | 22 | 24
participants | 14 | 18

2. Secondary Outcome: Cardiac Autonomic Neuropathy (CAN)
Description: Group differences in E/I ratio, a measure of cardiac autonomic function.
Time Frame: 18 months
Measure: Mean (Standard Deviation); unit: unit-less measure
Arm/Group | Exenatide | Glargine
Number analyzed (Participants) | 19 | 24
unit-less measure | 1.1 (0.1) | 1.1 (0.4)

3. Secondary Outcome: Cardiac Autonomic Neuropathy
Description: resting heart rate as marker of autonomic function at rest
Time Frame: 18 month
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Exenatide | Glargine
Number analyzed (Participants) | 19 | 24
beats per minute | 70 (9) | 77 (10)

4. Other Pre Specified Outcome: Intra-epidermal Nerve Fiber Density
Description: Exploratory endpoint: Regeneration of intra-epidermal nerve fibers after denervation by capsiacin.
Time Frame: 12 months
Population: Subset of study population
Measure: Mean (Standard Deviation); unit: nerve fibers per mm of skin
Arm/Group | Exenatide | Glargine
Number analyzed (Participants) | 11 | 11
nerve fibers per mm of skin | 2.1 (3.5) | 4.6 (2.9)

ADVERSE EVENTS:
Time Frame: From Screening to Study End: 1 year 7 months
Arm/Group | Exenatide | Glargine
Serious Adverse Events (participants affected / at risk) | 6/22 | 8/24
Other Adverse Events (participants affected / at risk) | 9/22 | 19/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exenatide (N=22) | Glargine (N=24)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Coronary Artery Bypass Graft (Cardiac disorders) | 0 (0) | 1 (1)
Congestive Heart Failure (Cardiac disorders) | 1 (1) | 1 (1) — Exacerbation of existing congestive heart failure
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Status Asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic Neuroendocrine Tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pregnancy (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholilithiasis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Thyroidectomy (Endocrine disorders) | 1 (1) | 0 (0)
Non-ST elevation myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Incarcerated Ventral Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
foot ulcer with cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Amputation of Toe (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — because of persistent cellulitis and non-healing ulcers
Bone Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) — 1 c-spine fracture due to motor vehicle accident 1 lower leg fracture because of fall
Severe Hypoglycemia (Endocrine disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exenatide (N=22) | Glargine (N=24)
Non-Serious Adverse Event (General disorders) | 9 (17) | 19 (39)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less